CLINICAL TRIAL: NCT06707181
Title: Comparative Study Between Silodosin , Tamsulosin , Silodosin Plus Tadalafil and Tamsulosin Plus Tadalafil As a Medical Expulsive Therapy for Lower Ureteral Stones
Brief Title: Comparative Study for Medical Therapy for Lower Ureteral Stones
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Hasnaa Osama, Lecturer at Clinical Pharmacy Department, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M713
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Lower Ureteral Stones
MeSH Terms: interventions — Tamsulosin; silodosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A (Active Comparator): Group A treated by silodosin 8mg.
  Interventions: Drug: • The study will include 180 randomly selected patients who met inclusion criteria were randomized into four groups: silodosin 8 mg (Group A), tamsulosin 0.4 mg (Group B), silodosin 8 mg plus tadalaf
- Group B (Active Comparator): Group B treated by a tamsulosin 0.4 mg .
  Interventions: Drug: • The study will include 180 randomly selected patients who met inclusion criteria were randomized into four groups: silodosin 8 mg (Group A), tamsulosin 0.4 mg (Group B), silodosin 8 mg plus tadalaf
- Group C (Active Comparator): Group C was treated with a combination of silodosin 8 mg and tadalafil 5 mg .
  Interventions: Drug: • The study will include 180 randomly selected patients who met inclusion criteria were randomized into four groups: silodosin 8 mg (Group A), tamsulosin 0.4 mg (Group B), silodosin 8 mg plus tadalaf
- Group D (Active Comparator): Group D treated by a combination of tamsulosin 0.4 mg and tadalafil 5 mg.
  Interventions: Drug: • The study will include 180 randomly selected patients who met inclusion criteria were randomized into four groups: silodosin 8 mg (Group A), tamsulosin 0.4 mg (Group B), silodosin 8 mg plus tadalaf

INTERVENTIONS:
Drug: • The study will include 180 randomly selected patients who met inclusion criteria were randomized into four groups: silodosin 8 mg (Group A), tamsulosin 0.4 mg (Group B), silodosin 8 mg plus tadalaf — • The study will include 180 randomly selected patients who met inclusion criteria were randomized into four groups: silodosin 8 mg (Group A), tamsulosin 0.4 mg (Group B), silodosin 8 mg plus tadalafil 5 mg (Group C) and tamsulosin 0.4 mg plus tadalafil 5 mg (Group D). Drugs are given for a maximal duration of 28 days.

SUMMARY:
The goal of this clinical trial is to compare the efficacy and adverse effects of different drugs as a medical expulsive therapy for lower ureteral stones. The main questions it aims to answer are:

* Which of the following are more effective silodosin, tamsulosin, silodosin plus tadalafil and tamsulosin plus tadalafil as a therapy for lower ureteral stones?
* What medical problems do participants have when taking these drugs?

Researchers will compare silodosin, tamsulosin, silodosin plus tadalafil and tamsulosin plus tadalafil to see which drug works better to treat lower ureteral stones Participants will:

* Take silodosin, tamsulosin, silodosin plus tadalafil or tamsulosin plus tadalafil every day for 28 days
* Visit the clinic once every 2 weeks for checkups and tests
* Keep a diary of their symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were adult patients aged 18 years and older with lower ureteral stones measuring 5-10 mm in diameter, diagnosed through imaging techniques such as kidney-ureter-bladder (KUB) x-rays or computed tomography (CT) scans.

Exclusion Criteria:

* Exclusion criteria included pregnant and lactating women, renal insufficiency, congenital urinary tract abnormalities, associated kidney stones or contralateral ureteric stones, solitary kidneys, associated infected stones, uncontrolled pain, severe hydronephrosis, history of allergy to the study medications and recent treatment for ureteral stones within the past 3 months (e.g., lithotripsy or surgery) .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-08-18 (Actual)

PRIMARY OUTCOMES:
Expulsion rate | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Fayoum University, Al Fayyum, Egypt